CLINICAL TRIAL: NCT05565534
Title: Optimizing Delivery of Diabetes Management During Breast Cancer Care
Brief Title: Diabetes Care for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-07025006; K01CA251645-01 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; PreDiabetes; Type 2 Diabetes
MeSH Terms: conditions — Breast Neoplasms; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study with non-randomized intervention and control groups. A nurse practitioner (NP) who is trained in diabetes on the oncology team will help manage diabetes for breast cancer patients undergoing cancer treatments. The control group will be enrolled first, followed by the experimental group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-practitioner led intervention group (Experimental): A nurse practitioner (NP) who is trained in diabetes on the oncology team will help manage diabetes for breast cancer patients undergoing cancer treatments
  Interventions: Behavioral: Nurse-practitioner led intervention
- Non-intervention (control) group (No Intervention): Patient will not have access to the nurse practitioner led intervention.

INTERVENTIONS:
Behavioral: Nurse-practitioner led intervention — * Face-to-face or virtual consultation with NP during chemotherapy infusion with individualized recommendations/medications AND patient education through the Patient Activated Learning System (PALS).
  * Weekly follow-ups from NP via phone, Zoom, or in-person (patient directed) for 12 weeks/course of chemotherapy.
  Arms: Nurse-practitioner led intervention group

SUMMARY:
The goal of this study is to find a new way to make diabetes care better for patients with breast cancer and diabetes who are currently receiving cancer treatment. We will have two groups, the researchers will decide who is in which group. One group will be working with a nurse who is trained in diabetes care while the other does not. This will allow the investigators to see if having a trained nurse as part of the care team can help improve the care the patients receive.

DETAILED DESCRIPTION:
The present study aims to develop a stakeholder-engaged nurse practitioner (NP)-led intervention to improve diabetes care for patients with breast cancer and diabetes who are undergoing cancer treatment.

This is a pilot feasibility study, in which we will use a quasi-experimental pre-post design with non-randomized intervention and control groups. In this feasibility study, the investigators will first enroll 38 eligible patients for the control group and collect effectiveness measures at baseline and follow-up (end of chemotherapy or other cancer treatment, ~12 weeks). Through chart review, the investigators will document cancer treatment regimen completion at follow-up. The investigators will then enroll 38 patients for the intervention group, collecting the effectiveness and implementation outcomes at the end of their treatment (~12 weeks).

The main hypothesis that will be tested in this pilot study is that a nurse practitioner embedded in the oncology team who is trained in diabetes management may successfully manage diabetes during active cancer care for patients undergoing cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed invasive cancer
* Plan to receive neo-adjuvant or adjuvant chemotherapy, targeted therapy, hormonal therapy, or radiation at Weill Cornell Medicine (WCM)

  * Age 18+ years
  * Pre-diabetes OR type 2 diabetes. Treatment with antidiabetic medication OR
* HbA1c greater than or equal to 5.7 OR
* Random glucose greater than or equal to OR
* Fasting blood glucose greater than or equal to 100

Exclusion Criteria:

* Patients receiving hospice care
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Recruitment Success Ratio | 2 years
  Number of participants recruited divided by the number of participants approached
Intervention Completion Success Ratio | 2 years
  Only for the interventional group The number of participants who completed intervention divided by the number of participants who enrolled
Data Collection Success Ratio | 2 years
  Number of participants who completed both surveys divided by the number of participants who were enrolled.
Patient Questionnaire: Self-report of intervention feasibility | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Feasibility of Intervention Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating that the intervention is very feasible, and lower scores (below 3) indicating the intervention is not feasible.
Provider Questionnaire: Self-report of intervention feasibility | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Feasibility of Intervention Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating that the intervention is very feasible, and lower scores (below 3) indicating the intervention is not feasible.
Patient Questionnaire: Self-report of intervention acceptability | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Acceptability of Intervention Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating more favorable attitudes toward the intervention and lower scores (below 3) indicating less favorable attitudes.
Provider Questionnaire: Self-report of intervention acceptability | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Acceptability of Intervention Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating more favorable attitudes toward the intervention and lower scores (below 3) indicating less favorable attitudes.
Patient Questionnaire: Self-report of intervention appropriateness | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Intervention Appropriateness Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating the intervention suits their needs well and lower scores (below 3) indicating the intervention does not fit their needs well.
Provider Questionnaire: Self-report of intervention appropriateness | Immediately post-intervention at the week 12 follow-up
  Questionnaire: Intervention Appropriateness Measure (4 items)
  Response Scale:
  For each item, respondents can choose a value from 1-5. Scales can be created for the measure by averaging responses for all 4 items for the overall score. The average score range is from 1 to 5 with higher scores indicating the intervention suits their needs well and lower scores (below 3) indicating the intervention does not fit their needs well.
Ratio of patients who receive a summary document at the end of the intervention | 2 years
  Number of patients who receive a summary document compared to the number of patients who complete the follow-up visit.
Number of in-person, virtual or phone contacts with the NP | 2 years
  This will assess the degree to which the intervention was implemented over the course of the study

SECONDARY OUTCOMES:
Change in Patient Self-report Responses of Diabetes Treatment Satisfaction Questionnaire | From baseline to week 12 follow-up visit
  Diabetes Treatment Satisfaction Questionnaire (8 items) DTSQ, score 0-36; higher scores reflecting higher satisfaction
Change in Patient Self-report Responses of Neuropathy as Measured By the PRO-CTCAE Survey | From baseline to week 12 follow-up visit
  PRO-CTCAE: Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events
  Neuropathy - PRO-CTCAE (2 items) 0-8 with higher scores representing worse neuropathy
Change in Patient Self-report Responses of Diabetes Distress Scale Questionnaire | From baseline to Week 12 follow-up
  Diabetes Distress Scale (17 items) A score of "1" indicates a particular item is not a problem or bother for the patient, whereas "6" represents an item is very concerning for the patient. To score, the patient's responses will be summed and then divided by the number of items in that scale. A mean score of 3 or higher (moderate distress) is considered as a level of distress that is above average.
Change in Patient Self-report Responses of the Audit of Diabetes Dependent QoL Questionnaire | From baseline to Week 12 follow-up
  Audit of Diabetes Dependent Quality of life (QoL) (15 items). For each item, respondents provide a score for both "impact" and "importance." Total weighted scores range from -9 to +3. Lower scores reflect poorer quality of life.
Change in Patient Self-report Responses of the Functional Assessment of Cancer Therapy-Breast Questionnaire | From baseline to Week 12 follow-up
  Functional Assessment of Cancer Therapy -Breast (44-items) measures quality of life for patients with breast cancer. Total scores range from 0-148 with higher scores representing better quality of life.
Change in number of Hospitalizations Since Cancer Diagnosis | From baseline to Week 12 follow-up
Change in number of Emergency Department (ED) Visits Since Cancer Diagnosis | From baseline to Week 12 follow-up
Number of missed chemotherapy doses | From baseline to Week 12 follow-up
  # of doses given subtracted from total # planned doses
Number of participants with a Delay in Chemotherapy Administration | From baseline to Week 12 follow-up
  # of days chemotherapy infusion was delayed from schedule date
Number of participants with Chemotherapy Dose Reductions | From baseline to Week 12 follow-up
  From the electronic medical chart: Indication if chemotherapy dose was reduced

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Pinheiro, PhD, MPH, Principal Investigator — Assistant Professor of Health Services Research in Medicine
Locations (3):
- United States (3):
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York-Presbyterian Queens, Flushing, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547

DOCUMENTS (1):
  • Informed Consent Form: Control Group (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT05565534/ICF_000.pdf